CLINICAL TRIAL: NCT06279702
Title: The Effect of First Aid Training on Knowledge, Skills and Motivation in Injuries Given to Secondary School Students With Serious Game Simulation and Comics
Brief Title: Serious Game Simulation and Comics in School Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ozlem Calisir, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OCalisir
Record Dates: First submitted 2024-02-09; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: First Aid
Keywords: serious game; first aid training; simulation

STUDY DESIGN:
Intervention Model Description: serious game and comics
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simulation group (Experimental): Students will be asked to perform first aid in the "First Aid Training for Injuries Serious Game Simulation Scenario without any first aid training and to fill in the data collection tools integrated into the game. Correct approach training to the injured will be given through "First Aid in Injuries Training Serious Game Simulation Scenario CORRECT PRACTICES TRAINING integrated into the serious game. Upon completion of the training, the next step will be free work time. Students will be able to play as many games as they want.
  Interventions: Other: SERIOUS GAME
- Comic Group (Experimental): Students will be given First Aid Training in Injuries, prepared in the form of a comic book.
  Interventions: Other: COMICS
- other (No Intervention): Training will not be provided within the scope of serious games and with comic books.

INTERVENTIONS:
Other: SERIOUS GAME — Students will play serious game that about first aid.
  Arms: simulation group
Other: COMICS — students will learn comics that about first aid.
  Arms: Comic Group

SUMMARY:
The aim of the study is to determine the effect of first aid training for injuries given to secondary school students through serious game simulation and comic books on knowledge, skills and motivation.

Hypotheses:

H1: First aid training given through simulation applications affects the level of knowledge.

H2: First aid training given through simulation applications affects the skill level.

H3: First aid training given with simulation application affects motivation.

H4: First aid training given with comics affects the level of knowledge.

H5: First aid training given with comic books affects the skill level.

H6: First aid training given with comics affects motivation.

METHOD: The research will be conducted as a randomized controlled experimental study with a pre-test-post-test design with children studying in the 5th and 6th grades of schools in the central district of Aksaray. One group will be given first aid training for injuries prepared with serious games, the other group will be given first aid training for injuries prepared with comic books. No intervention will be made to the control group. Serious game scenario software prepared based on the literature will be integrated into the computer. Appropriate statistics will be made after the research by applying the prepared data collection tools. With this research, the gap in the literature will be filled, children's first aid knowledge and skills in injuries will be increased, and school health nurses will be provided with up-to-date teaching material.

DETAILED DESCRIPTION:
Accidents are one of the leading causes of death in children and adults and threaten health on a global scale. Exposure is especially high during childhood. Lost human resources due to premature deaths and large health care costs due to disabled individuals impose a serious burden on countries. This burden puts the growth rate, welfare, and productivity of countries at risk. First aid is provided throughout the country to prevent the development of such risks.

The practices must be carried out actively. The long-term impact of first aid interventions based on knowledge and skills is proportional to the training provided. For training to be effective and permanent, it may be more effective to use materials/methods brought by developing technology. It is thought that first aid training given through serious game simulation will also be effective. These serious games, accessed via computers, will provide students with plenty of experience with both ease of use and repetitive practice. It is known that emergencies requiring first aid can cause panic. Being calm when responding to an injured person can only be improved through experience. A realistic virtual environment designed with serious games can be effective in gaining experience. The designed serious game simulation teaching material can be applied in all schools across the country. First aid can also be prepared for all issues other than injuries. Thus, a teaching material that can affect large audiences will be developed.

The research will be conducted as a randomized controlled experimental study with a pre-test post-test design.

The research will be conducted with children studying in the 5th and 6th grades of schools in the central district of Aksaray, affiliated with the Ministry of National Education (MEB) of the Republic of Turkey.

The population of the research consists of 21,343 (public + private) children studying in primary (secondary) institutions in Aksaray. Of these students, 5440 students are in the 5th grade and 5277 students are in the 6th grade.

In the research, with statistical support, the sample size was used using G*Power 3.1.9.7, the power of the study was calculated as 95% confidence level, the effect size was 0.25, the alpha value was 0.05, and the sample number was 54 (simulation group 18, comic book group 18, control group 18) students.

ELIGIBILITY:
Inclusion Criteria:

* Secondary schools with computer laboratories,
* 5th and 6th-grade secondary school students whose families gave permission and volunteered to participate in the research,
* Not an inclusion student,
* No physical or mental disability or limb loss,
* Able to understand, speak, and write Turkish,
* Students who have not taken courses on first aid.

Exclusion Criteria:

* Students who have not completed all stages of the education program,
* Students whose parents or themselves wish to withdraw from the study will be removed from the study groups.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
Motivation Scale for Teaching Materials | The measurement will start 15 minutes before the serious game, comics and will end 15 minutes after the serious game, comics.
  It is stated that the highest score that can be obtained from the scale is 165 and the lowest score is 33. High total score It means that students' motivation levels regarding the teaching material are high.
Student Knowledge Level Evaluation Form for First Aid Application in Injuries | The measurement will start 15 minutes before the serious game, comics and will end 15 minutes after the serious game, comics.
  It was prepared by researchers in line with the literature.The form consists of a total of 19 questions to which students can answer "True" or "False".
Student Skill Level Evaluation Form for First Aid Application in Injuries | While students intervene in the serious game, this form will be filled automatically by the serious game software.
  It was prepared by researchers in line with the literature and it consists of 13 items.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çalışır, pHD, Principal Investigator — TC Erciyes University
Locations (1):
- Özlem Çalışır, Aksaray, Center, Turkey (Türkiye)